CLINICAL TRIAL: NCT07238049
Title: READ-OUT - REAl World Dementia OUTcomes: Observational Study
Brief Title: REAl World Dementia OUTcomes: Observational Study
Acronym: READ-OUT
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Cambridge (Other); University of Edinburgh (Other); Greater Manchester Mental Health NHS Foundation Trust (Other); University of Bristol (Other); Queen Mary University of London (Other); West London NHS Trust (Other); University College, London (Other); Imperial College London (Other); Aneurin Bevan University Health Board (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: 24/WA/0330; ARUK-BBC2023-001 (Other Grant/Funding Number: Alzheimer's Research UK)
Record Dates: First submitted 2025-09-01; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease (AD); Mild Cognitive Impairment (MCI); Dementia
Keywords: Dementia; Blood-based biomarkers; Diagnosis; Cognitive impairment; memory clinics
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples With DNA — Blood samples (serum and plasma) will be retained for biomarker analysis and future research. DNA will be extracted for genotyping using whole genome enzymatic methylation sequencing with 30-50x coverage on Illumina NovaSeq X+. Cell-free DNA will be analysed using contemporary bioinformatics pipelines integrating multiple analytical approaches. Samples will be stored in the biorepository for exploratory biomarker development and future research with appropriate consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
READ-OUT observational study will investigate blood-based biomarkers for dementia in real-world clinical settings. This 3-year observational study will include 3165 people, males or females aged 45 years or older, with cognitive impairment of any severity.

Participants provide blood samples and complete questionnaires about quality of life and healthcare use, with some having additional follow-ups at 2 weeks and 1 year. The study will assess reliability and accuracy of blood tests in diagnosing dementia.

DETAILED DESCRIPTION:
Dementia affects a growing number of people in the UK, with significant costs for individuals, families, and society. There is an urgent need for accurate diagnosis of dementia to allow early intervention and support when people can still make decisions about their care.

Current dementia diagnosis in memory clinics relies on clinical assessment, cognitive testing, and brain scans (MRI or CT). Only a small proportion of UK patients have access to more specific tests like PET brain scans or spinal fluid analysis, which are expensive and not widely available.

Recent developments have shown that blood tests can accurately detect the underlying brain changes of dementia, particularly Alzheimer's disease. In research studies, these blood-based biomarkers (ptau217, AB42/40 ratio, GFAP, NFL etc) have successfully identified people with Alzheimer's disease when compared to clinical diagnoses, gold standard brain scans, and post-mortem brain examination. These blood tests also show promise for predicting people with future dementia risk.

However, most research has been conducted in younger, less diverse populations than those seen in real-world memory services. Blood-based biomarkers are not yet used in routine NHS practice, and more work is needed to test how well they perform in representative UK populations. We also need to understand whether people want to know their blood test results, what information they want, and how this is best communicated.

The READ-OUT study will test blood-based biomarkers in people attending memory clinics across the UK (30 NHS sites), ensuring participants represent the full diversity of people with dementia or memory concerns (30% from underrepresented groups). Participants will provide a 40ml blood sample and complete questionnaires about quality of life, healthcare use, and attitudes toward blood testing for dementia. The accuracy of blood biomarkers will be compared against established diagnostic methods including expert clinical review, brain scans, spinal fluid tests, and long-term health record follow-up.

The study includes three optional sub-studies: test-retest reliability of blood biomarkers (10% of participants returning after 1-2 weeks), investigating disease progression over one year (20% of participants), and evaluating whether people can collect blood samples at home using finger-prick cards (75 participants).

The study will determine which blood biomarkers are most accurate for diagnosing different types of dementia, predict disease progression, and assess their cost-effectiveness in the healthcare system. Results will inform whether these tests should be integrated into NHS clinical pathways and will guide the design of READ-OUT Phase 2, a randomized trial testing whether providing blood biomarker results to patients and doctors improves clinical care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

The participant may enter the study if ALL of the following apply:

* Willing and able to give informed consent for participation in the study (translation needs for study information and forms for non-English speakers will be defined locally) OR Adults who otherwise lack the capacity to consent but for whom advice regarding participation has been obtained via a consultee using the personal or nominated consultee process
* Male or Female, aged 45 years and above
* Referred or referable with cognitive or behavioural symptoms and/or diagnosed with a cognition related disorder; including those with subjective cognitive impairment and functional disorders.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Lack of venous access
* Unwilling to consent to NHS data linkage or in Northern Ireland, unwilling to allow long term follow up by access to electronic NHS records.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People referred to, eligible for referral or already under review at primary and/or secondary memory assessment services (including memory clinics, brain health clinics) with some form of cognitive symptoms and/or cognitive disorders of any severity will be eligible for recruitment. Also, we recruit a subset of individuals who are not under a secondary care memory clinic but who have a clinical picture that would be suitable for secondary care assessment in memory clinic services.
Sampling Method: Non-Probability Sample
Enrollment: 3165 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of blood-based biomarkers for dementia diagnosis | baseline and at 52 weeks
  Accuracy, Positive and Negative predictive value in regard to diagnosis and, where available, gold standard biomarker measures (clinical consensus, cerebrospinal fluid, CSF, positron emission tomography, PET)
Feasibility and acceptability of blood-based biomarkers for dementia diagnosis | baseline, at 2 weeks and 52 weeks
  Recruitment metrics at site level Acceptability patient questionnaires Patient and Public Involvement qualitative data around acceptability of BBM collection
Cost-effectiveness of blood biomarkers in a real-world cognitive disorders population | baseline and at 52 weeks
  Health-related quality of life (HR-QoL) Healthcare utilisation

SECONDARY OUTCOMES:
Disease prediction utility of blood-based biomarkers in diverse cognitive disorders populations | baseline and at 52 weeks
  Cognitive score progression, MCI to dementia conversion, Institutionalisation, or Death, ethnicity.
Optimal individual or sets of biomarkers for separate dementia aetiologies | baseline, at 2 weeks and 52 weeks
  Accuracy, Positive and Negative predictive value in regard to subgroups of dementia diagnosis
Impact of sample processing delays on the accuracy of blood biomarkers | Baseline study visit
  BBM levels obtained from samples of varying degrees of processing delays
The test-retest reliability of blood biomarkers | Baseline study visit, 1-2 week visit
  BBM levels obtained from repeated sampling at baseline and after 1-2 week - a sub- study involving 10% of the participant sample.
  Whether samples taken at different time points are comparable will be assessed
The utility of remote blood test kits | Baseline study visit
  Comparison of BBM levels obtained from phlebotomy and blood spot cards/Capillary Tubes involving 75 individuals within the sample; Accuracy, positive and negative predictive value for blood spot card/Capillary Tubes BBMs
Understanding participant preferences on disclosure of biomarker status in dementia diagnosis | baseline and at 52 weeks
  Evaluation of participants' views on what information they wish to receive about their biomarker status, the preferred timing of disclosure, and the most appropriate method of communication. Quantitative data will be collected via questionnaires completed by all participants at baseline. A qualitative sub-study involving 15-20 participants, supported by the trial PPIE group, will explore experiences and preferences in greater depth through interviews and/or focus groups.

OTHER OUTCOMES:
Exploratory analysis to support development of novel multi-omics assays for dementia diagnosis and prognosis | baseline and at 52 weeks
  Exploratory analyses will focus on identifying and validating potential diagnostic or prognostic biomarkers through multi-omics approaches

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Raymont, Principal Investigator — University of Oxford
Locations (27):
- United Kingdom (27):
  - Betsi Cadwaladr University Health Board, Bangor
  - ReMind UK, Bath
  - Belfast Health & Social Care Trust, Belfast
  - Dorset HealthCare University NHS Foundation Trust, Bournemouth
  - Berkshire Healthcare NHS Foundation Trust, Bracknell
  - Bradford District Care NHS Foundation Trust, Bradford
  - North Bristol NHS Trust, Bristol
  - Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge
  - Devon Partnership NHS Trust, Exeter
  - Barts Health NHS Trust, London
  - East London NHS Foundation Trust, London
  - South London and Maudsley (SLaM), London
  - St George's Hospital, London
  - West London NHS Trust, London
  - Greater Manchester Mental Health Foundation Trust, Manchester
  - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne
  - Aneurin Bevan University Health Board, Newport
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Health NHS Trust, Oxford
  - Lancashire & South Cumbria NHS Foundation Trust, Preston
  - Surrey and Borders Partnership NHS Foundation Trust, Redhill
  - Sheffield Health and Social Care NHS Foundation Trust, Sheffield
  - Sheffield Teaching Hospital, Sheffield
  - Hampshire and Isle of Wight NHS Foundation Trust, Southampton
  - University Hospital Southampton, Southampton
  - Midlands Partnership University NHS Foundation Trust, Stafford
  - Sussex Partnership NHS Foundation Trust, Worthing

IPD SHARING:
Plan to Share IPD: Yes
Anonymised (linked) BBM and genetic data will be available for access (not copying/export) via the DPUK Data Portal (https://portal.dementiasplatform.uk/) upon an approved data/sample access proposal. It offers a secure, fully auditable data repository (currently facilitating access to data for over 3.6m individuals across more than 60 cohorts). A curated (standardised/harmonised) dataset will be made available to eligible researchers within the DPUK Trusted Research Environment (TRE) which is at the core of the Data Portal.
URL: https://portal.dementiasplatform.uk/